CLINICAL TRIAL: NCT07261683
Title: A Phase II Study Evaluating the Efficacy and Safety of Weekly Paclitaxel or Nab-Paclitaxel Combined With Pembrolizumab and Mirabegron in Patients With Recurrent Ovarian Cancer
Brief Title: Phase II Study of Weekly Paclitaxel/Nab-Paclitaxel, Pembrolizumab, and Mirabegron for Recurrent Ovarian Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Obstetrics & Gynecology Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Xin Wu, Director, Obstetrics & Gynecology Hospital of Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUOBGY-2025-202
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Cancer; Immunotherapy; Pembrolizumab
Keywords: ovarian cancer; immunotherapy
MeSH Terms: conditions — Ovarian Neoplasms | interventions — pembrolizumab; mirabegron

STUDY DESIGN:
Masking Description: This is a single-arm, open-label, Phase II interventional study designed to evaluate the efficacy and safety of weekly paclitaxel or nab-paclitaxel in combination with pembrolizumab and mirabegron in patients with recurrent ovarian cancer. All eligible participants will receive the same treatment regimen without randomization or masking. The study aims to assess treatment response, safety profile, and preliminary clinical benefit in this target population.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Weekly Paclitaxel/Nab-Paclitaxel, Pembrolizumab, and Mirabegron (Experimental): Participants receive weekly paclitaxel/nab-paclitaxel plus pembrolizumab via intravenous (IV) infusion plus on Day 1 of each 21-day cycle orally with daily mirabegron until intolerance or disease progression.
  Interventions: Drug: Weekly Paclitaxel/Nab-Paclitaxel, Pembrolizumab, and Mirabegron

INTERVENTIONS:
Drug: Weekly Paclitaxel/Nab-Paclitaxel, Pembrolizumab, and Mirabegron — Participants receive weekly paclitaxel/nab-paclitaxel plus pembrolizumab via intravenous (IV) infusion plus on Day 1 of each 21-day cycle orally with daily mirabegron until intolerance or disease progression.

SUMMARY:
The goal of this clinical trial is to learn if drug regimen weekly paclitaxel/nab-paclitaxel, pembrolizumab, and mirabegron works to treat relapsed ovarian cancer in adults. It will also learn about the safety of the drug regimen. The main questions it aims to answer are:

i) Does drug weekly paclitaxel/nab-paclitaxel, pembrolizumab, and mirabegron reduce tumor volume? ii) What medical problems do participants have when taking drug weekly paclitaxel/nab-paclitaxel, pembrolizumab, and mirabegron?

Participants will:

i) Take drug paclitaxel/nab-paclitaxel every week and pembrolizumab every 21 days with everyday mirabegron ii) Visit the clinic once every 2 months for checkups and tests iii) Keep a diary of their symptoms

ELIGIBILITY:
Inclusion Criteria:

* Has provided documented informed consent for the study.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Has histologically confirmed epithelial ovarian, fallopian tube, or primary peritoneal carcinoma.
* Has received a front line platinum-based regimen (administered via either intravenous or intraperitoneal route) per local standard of care or treatment guideline following the primary or interval debulking surgery with documented disease recurrence (note: Maintenance treatment following the front line treatment is permitted and counted together as part of the front line treatment).
* Has a platinum-free interval (PFI) of < 12 months if the last regimen received is a platinum-based, or a treatment-free interval (TFI) of < 12 months if the last regimen received is a non-platinum-based.
* Has measurable disease at baseline based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Has a life expectancy of ≥12 weeks.
* Has provided a tumor tissue sample either collected from prior cytoreductive surgery or fresh newly obtained tumor tissue at screening.
* Has adequate organ function.
* Has not recovered from AEs to ≤ Grade 1 or prior treatment level due to a previously administered agent.

Exclusion Criteria:

* Has nonepithelial cancers, borderline tumors, mucinous, seromucinous that is predominantly mucinous, malignant Brenner's tumor and undifferentiated carcinoma.
* Has received prior therapy with an anti-programmed cell death (PD)-1, anti-PD-L1, anti-PD-L2 agent or with an agent directed to another co-inhibitory T-cell receptor (e.g. cytotoxic T-lymphocyte-associated antigen-4 [CTLA-4], tumor necrosis factor receptors OX-40 or CD137).
* Has received prior systemic anticancer therapy including radiation therapy or maintenance therapy within 4 weeks before enrollment.
* Has severe hypersensitivity (≥Grade 3) or uncontrolled hypertension to paclitaxel/nab-paclitaxel, pembrolizumab, mirabegron and any of their excipients.
* Has undergone major surgery within 3 weeks before enrollment or has complications/sequelae that have not yet recovered.
* Has a known additional malignancy that progressed or required active treatment within the last 5 years.
* Is pregnant or breastfeeding.
* Has a history of allogenic tissue/solid organ transplant.
* Has a history of thrombotic disorders, hemorrhage, hemoptysis, or active gastrointestinal bleeding within 6 months before enrollment.
* Has a history of active autoimmune disease.
* Has an active infection requiring systemic therapy.
* Has a history of human immunodeficiency virus (HIV) infection.
* Has a history of Hepatitis B or C virus infection.
* Has a history or current evidence of any condition, therapy, laboratory abnormality, or other circumstance that might confound the results of the study.
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligible participants must self-identify as female and have a diagnosis of ovarian cancer with current or historical ovarian tissue.
Enrollment: 20 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Month 6
  Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by Blinded Independent Central Review (BICR). ORR was defined as the percentage of participants who had a Complete Response (Disappearance of all target lesions) or a Partial Response (≥30% decrease in the sum of the longest diameter of target lesions) using RECIST 1.1 based on BICR.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) at 6 Months | Month 6
  PFS was defined as the time from first dose of study treatment to the first documented progressive disease (PD) per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm.
  The appearance of ≥1 new lesion is also PD. PFS at 6 months is defined as the percentage of patient who was progression free at 6 months from the date of first study treatment.
Overall Survival (OS) at 6 Months | Month 6
  OS at 6 months is defined as the percentage of patients who are alive at 6 months from the date of first study treatment.
Progression Free Survival (PFS) at 12 Months | Month 12
  PFS was defined as the time from first dose of study treatment to the first documented progressive disease (PD) per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and an absolute SOD increase of ≥5 mm.
  The appearance of ≥1 new lesion is also PD. PFS at 12 months is defined as the percentage of patient who was progression free at 12 months from the date of first study treatment.
Overall Survival (OS) at 12 Months | Month 12
  OS at 12 months is defined as the percentage of patients who are alive at 12 months from the date of first study treatment.
Incidence of grade 3-4 Adverse Events (AEs) | up to 1 month after the end of treatment
  Incidence of grade 3-4 AEs, according to CTCAE, version 5.0

OTHER OUTCOMES:
Exploratory outcome: biomarkers testing and efficacy of anti-tumor immunity | Baseline and 6 months from the the date of first study treatment
  Biomarker testing for PD-L1 expression in exploratory analysis.
Exploratory outcome: biomarkers testing and efficacy of anti-tumor immunity | Baseline and 6 months from the the date of first study treatment
  Biomarker testing for BMI (weight and height will be combined to report BMI in kg/m^2) in exploratory analysis.
Exploratory outcome: biomarkers testing and efficacy of anti-tumor immunity | Baseline and 6 months from the the date of first study treatment
  Biomarker testing for tumor microenvironment (including density and state of CD8+ T cells density and other immune cells) in exploratory analysis.
Exploratory outcome: biomarkers testing and efficacy of anti-tumor immunity | Baseline and 6 months from the the date of first study treatment
  Biomarker testing for circulating anti-tumor immunity (including density and state of CD8+ T cells density and other immune cells) in exploratory analysis.
Exploratory outcome: biomarkers testing and efficacy of anti-tumor immunity | Baseline and 6 months from the the date of first study treatment
  Biomarker testing for transcriptome in exploratory analysis.
Exploratory outcome: biomarkers testing and efficacy of anti-tumor immunity | Baseline and 6 months from the the date of first study treatment
  Biomarker testing for genome in exploratory analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Obstetrics and Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No